CLINICAL TRIAL: NCT05734859
Title: A Pilot Study of Drinking Electrolyzed Hydrogen-rich Alkaline Reduced Water Generated by Alkaline Ionizer (BTM-1200) on the Chronic Functional Constipation
Brief Title: Drinking Effect of Electrolyzed Alkaline Reduced Water on Functional Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wonju Severance Christian Hospital (Other)
Responsible Party: Principal Investigator, Kyu Jae Lee, Professor, Wonju Severance Christian Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMB-2022-03
Record Dates: First submitted 2023-01-26; First posted 2023-02-21 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Chronic Constipation
Keywords: constipation; hydrogen-rich alkaline ionized water; complete spontaneous bowel movement; patient assessment of constipation-symptoms; patient assessment of constipation-quality of life
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Intervention Model Description: comparison between baseline and post-treatment in single group
Masking Description: No need of blinding
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EHARW Treatment group (Experimental): The experimental group will drink a total amount of 20 mL/ kg body weight/day of EHARW for 4 weeks on an empty stomach according to the researcher's instruction.
  Interventions: Device: Electrolyzed Alkaline Ionizer

INTERVENTIONS:
Device: Electrolyzed Alkaline Ionizer — Patients will drink EHARW calculated by 20 mL/kg body weight/day which can be divided into several times a day for drinking. The patient is recommended to drink water in an empty stomach and to drink water generated from the device as soon as possible.
  Other Names: BTM-1200

SUMMARY:
The goal of this clinical trial is to investigate drinking effect of electrolyzed hydrogen-rich alkaline reduced water (EHARW) in chronic constipation patients. The main question is that drinking EHARW will improve the symptoms of chronic constipation for 4 weeks.

Participants will drink EHARW (20 mL/kg of body weight/day) generated from the experimental device for 4 weeks.

DETAILED DESCRIPTION:
Patients diagnosed with constipation will be recruited and screened according to the inclusion and exclusion criteria after sign in the informed consent form. The selected patients will be enrolled. The experimental device (BTM-1200, Bion-Tech, Gyeonggi-do, Korea) will be installed at each patient's house. The researcher will instruct patients drinking method. The patients will drink a total of 20 mL/kg of body weight/day of EHARW (pH 9.5) in 3-different times, and drink directly from the device on an empty stomach for 4 weeks. The clinical trial is conducted in a single group without a control group, and the efficacy is evaluated by comparing the symptoms of constipation pre- and post-intervention. The primary outcome is the proportion of responders based on frequency of complete complete spontaneous bowel movement (CSBM).

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 19 to 70 years old
* Those who meet the criteria for Roma Ⅳ function constipation
* Symptoms begin before 6 months and last for more than 3 months
* Those who do not have organic lesions that may cause constipation
* A patient who has personally signed the consent form
* If all the criteria meet

Exclusion Criteria:

* Those taking drugs such as opioid analgesics, antipsychotics, calcium blockers, and parasympathetic antagonists
* Kidney disease (renal failure, potassium excretion disorder, etc.)
* Patients with colon-related diseases (colon cancer, intestinal stenosis, rectal flow, anal fissure, rectal bleeding), diabetes, thyroid dysfunction, or anemia
* Pregnant or lactating women
* In addition to the above, those who are judged to be difficult to conduct research by the clinical trial director
* Excluded if at least one of the above criteria meet

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-11-30 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2023-01-13 (Actual)

PRIMARY OUTCOMES:
Complete spontaneous bowel movement (CSBM) frequency | 4 weeks treatment
  CSBM is used to access the frequency of bowel movement. This indicates the efficacy of EHARW (pH 9.5) after 4-weeks of treatment in chronic constipation patients.

SECONDARY OUTCOMES:
Bristol stool scale score | 4 weeks treatment
  Fecal form is accessed by using Bristol stool scale. Fecal form indicate hardness of stool. Higher score present improvement of constipation symptoms. Similarly other questionnaires using self observation diary was also assessed including straining at defecation, stiffness of the stool, sensation of incomplete evacuation, and sensation of obstruction.
Patient assessment of constipation-symptoms (PAC-SYM) Questionnaire | 4 weeks treatment
  PAC-SYM is used to access constipation symptoms of patient before and after the intervention. This tool is categorized into 3 (abdominal, rectal, stool), and includes total 12 questions. Higher score present improvement of constipation symptoms.
Patient assessment of constipation-quality of life (PAC-QOL) Questionnaire | 4 weeks treatment
  PAC-QOL is used to access constipation-related quality of life before and after the intervention. This tool is categorized into 4: physical discomfort, psychological discomfort, worries and satisfaction, and consists of 28 questions. Higher score present improvement of constipation symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Kyu-Jae Lee, Ph.D., Principal Investigator — Department of Convergence Medicine, Wonju College of Medicine, Yonsei University
Locations (1):
- Wonju College of Medicine, Wŏnju, Ganwon-do, South Korea

IPD SHARING:
Plan to Share IPD: No